CLINICAL TRIAL: NCT03078530
Title: Probiotic (Visbiome) for Gulf War Illness
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ashok Tuteja (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ashok Tuteja, Professor Gastroenterology, VA Salt Lake City Health Care System
Organization: VA Salt Lake City Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00059006
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Gulf War Illness
Keywords: GWI; IBS; Irritable Bowel Syndrome; Gulf War Illness; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo (not an active drug/ Inactive component) is given to this group
  Interventions: Drug: Placebo
- Visbiome (Experimental): Visbiome (probiotic mixture) is given to this group.
  Interventions: Drug: Visbiome
- VSL #3 (Experimental): VSL #3 (probiotic mixture) is given to this group
  Interventions: Drug: VSL#3

INTERVENTIONS:
Drug: Placebo — This is a pill with inactive ingredients
  Other Names: Placebo/ Sugar pill
  Arms: Placebo
Drug: Visbiome — This is a probiotic mixture available to randomized study participants, starting with subject 29
  Arms: Visbiome
Drug: VSL#3 — This is a probiotic mixture available to the first 28 subjects randomized to the study
  Arms: VSL #3

SUMMARY:
The overall objective is to determine whether Visbiome will improve

1. intestinal symptoms of Irritable Bowel Syndrome (IBS) and
2. non-intestinal symptoms (fatigue, joint pain, insomnia, general stiffness and headache) associated with IBS. All of these symptoms are part of the Gulf War (GW) illness.

DETAILED DESCRIPTION:
Specific Aims:

Aim # 1: Determine the efficacy of Visbiome on IBS symptoms in GW veterans.

Hypothesis: Treatment with Visbiome compared to placebo will improve global and individual symptoms of IBS

Aim #2 Determine the efficacy Visbiome in reducing non-intestinal symptoms of IBS (fatigue, joint pain, insomnia, general stiffness and headache).

Hypothesis: Treatment with Visbiome compared to placebo will improve non-intestinal symptoms of IBS in GW veterans.

Aim #3 Determine whether changes in gut flora and plasma cytokines correlate with treatment response in GW veterans

ELIGIBILITY:
Inclusion Criteria:

1. First GW veterans, Men and women age 35-75 years,
2. Rome III criteria for IBS and two or more of the non-intestinal symptoms (chronic-once a week or more often-fatigue, joint pains, insomnia, general stiffness, and headache)
3. Symptoms of > 6 months duration,
4. No significant findings on physical examination, Complete Blood Count (CBC) and clinical chemistry panel.
5. Normal gross appearance of the colonic mucosa other than erythema and polyps
6. Negative Tissue transglutaminase (TTG) for celiac disease,
7. Normal thyroid function.
8. Veterans with psychological disorders will not be excluded but will be identified for sub-group analysis.
9. Stable medication regimen for more than a month

Exclusion Criteria:

1. Current evidence of any lower gastrointestinal disorder such as celiac disease or inflammatory bowel disease
2. History of/or presence of systemic malignancy (patients with skin and other cancers in remission for more than 5 years are allowed in the study
3. Clinically significant chronic disease: HIV, cardiac, pulmonary, hepatic or renal dysfunction.
4. Presence of Giardia antigen, and Clostridium difficile toxin in stool,
5. Abnormal blood test for thyroid stimulating hormone, tissue transglutaminase antibody
6. Current effects of drug or alcohol abuse
7. Investigator perception of patient's inability to comply with study protocol
8. Recent change in gastrointestinal medications
9. Use of any antibiotic in the last 1 months
10. Positive pregnancy test
11. Subject is currently participating in another research protocol that could interfere or influence the outcome measures of the present study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09-13 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in the bowel symptom scale from the baseline | Baseline to 8 weeks
  Efficacy of Visbiome in IBS related symptoms in GW illness is measured using BSS at 8 weeks

SECONDARY OUTCOMES:
Change in chronic fatigue (1-5 scale) from baseline | baseline to 4 weeks
  Efficacy of Visbiome in reducing non-intestinal symptoms of IBS is measured using chronic fatigue scale at 4 weeks.
Change in chronic fatigue (1-5 scale) from baseline | baseline to 8 weeks
  Efficacy of Visbiome in reducing non-intestinal symptoms of IBS is measured using chronic fatigue scale at 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Tuteja, MD, MPH, Principal Investigator — George E Wahlen VA Medical Center
Locations (1):
- George E Wahlen VA Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No